CLINICAL TRIAL: NCT02991391
Title: Expansion of the COPD At-risk Module in 4 States BRFSS Telephone Health Surveys
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Wake Forest University Health Sciences (Other); Medical University of South Carolina (Other); University of Kentucky (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00059852
Record Dates: First submitted 2016-10-06; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: COPD; Respiratory Symptoms; Tobacco Use; Asthma; Disparities; Air Quality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Signs and Symptoms, Respiratory; Tobacco Use; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: None, use of a questionnaire — Telephone health survey using 2015 Behavioral Risk Factor Surveillance Survey in Texas, Florida, South Carolina, and Kentucky that includes questions regarding tobacco exposure and respiratory symptoms

SUMMARY:
This cross-sectional survey study is intended to describe the characteristics of adults in 4 US states with regards to respiratory symptoms and tobacco exposure, utilizing an existing state-administered, CDC overseen Behavioral Risk Factor Surveillance System telephone health survey. The primary goal of study is to describe the sociodemographics, health behaviors, and presence of chronic diseases in persons with or at risk of having chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to determine the prevalence and health-related characteristics of adults who are at high risk for COPD, but have never been diagnosed. The second objective of this study is to determine the frequency and type of respiratory symptoms in the general adult population among 4 states. The third objective is to describe respiratory symptoms in the adult population in relationship to other chronic diseases such as COPD, asthma, obesity and others. The fourth objective is to engage other states to add the Module into their BRFSS as early as 2017 to aid in efforts to decrease the burden of COPD.

Procedures: The COPD At-risk Module will be incorporated into 4 state's 2015 BRFSS telephone health survey (SC, TX, FL, and KY). The COPD At-Risk Module was derived from previously published COPD case-finding and population screening questionnaires. The 4 questions contained in the Module are: 1) How many years have you smoked tobacco products? (asked of those that say they smoked > 100 cigarettes/lifetime, which is part of core survey), 2) In the last 30 days, how often are you short of breath? 3) How often do you cough up mucus or phlegm? and 4) In the last 12 months, to what extent would you say your physical activities are limited by shortness of breath? One additional question, age in years, is already contained in the BRFSS, and when combined with the other 4 questions, will allow estimation of survey participant's risk of COPD. The COPD risk categories are: 1) diagnosed COPD (self-report of provider diagnosis of COPD), 2) high risk for COPD (self-report of frequent respiratory symptoms based on participant responses plus at least 10 years of tobacco product use), and 3) low risk (neither diagnosed COPD or in high-risk group).

Each state's BRFSS group (state government epidemiology departments) will undertake the BRFSS telephone survey beginning January 2015 as part its normal annual state-based health surveillance. The core BRFSS survey has been developed by the CDC and minor changes in the core survey may occur each year. Individual states often have additional state-specific questions such as those requested by outside organizations or individuals, such as done with this study. The study investigators have requested and received approval to add the "COPD at-risk Module" that consists of 4 questions will be added to the 70-plus sociodemographic and health characteristic questions already included in the BRFSS.

Per CDC guidelines, potential survey respondents may refuse to participate or answer any question in the survey. Using a scripted BRFSS, trained interviewers will collect data using an independent prob¬ability sample of households through landline and cellular telephones of non-institutionalized persons. Based on past BRFSS surveys, the participant response rates have declined from ~ 60% to ~ 50% due to inclusion of cell phones along with landlines beginning in 2011. According to the CDC, the inclusion of cell phones and landline phones better represents the general adult population, especially in younger adults. A detailed description of the survey's design and random sampling procedures is available in the BRFSS Policies, Procedures, and Protocol Document, 2013 . The BRFSS has been approved as exempt research by the CDC's institutional review board.

Study Population It is projected that there will be ~ 45,000 non-institutionalized adults (> 18 years) who will complete the 2015 BRFSS telephone health survey among the 4 participating states - KY, SC, TX, and FL. These 4 states represent a significant segment of the COPD population in the US based upon prior COPD prevalence estimates and COPD-related hospitalizations among Medicare recipients. Of note, Kentucky has the highest prevalence of COPD in the US. For each state, cell phone and landline phones are randomly selected based on pre-determined goals for geographics and socio-demographics per state and CDC procedures. Hispanics can also participate in the telephone survey through interpreters. Only one adult in each household that is contacted can complete the survey. Of all potential survey respondents, about one-half will provide complete data for the telephone survey.

Data Collection and Confidentiality Collection of survey data from participants will start January 2, 2015 and be completed by the end of 2015. Prior to states analyzing and releasing survey data in 2016, the CDC will undertake an internal review of each state's survey data by May 2016.

Data files from the states and CDC that are shared with outside investigators contain no PHI. After states review and analyze their survey data, it is then available to be released to the public upon request, this includes investigators of this study.

ELIGIBILITY:
Inclusion Criteria:

* willingness to complete telephone health survey

Exclusion Criteria:

* unwillingness to compete telephone health survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is projected that there will be ~ 50,000 non-institutionalized adults (> 18 years) who will complete the 2015 BRFSS telephone health survey among the 4 participating states - KY, SC, TX, and FL. These 4 states represent a significant segment of the COPD population in the US based upon prior COPD prevalence estimates and COPD-related hospitalizations among Medicare recipients. Of note, Kentucky has the highest prevalence of COPD in the US. For each state, cell phone and landline phones are randomly selected based on pre-determined goals for geographics and socio-demographics per state and CDC procedures. Hispanics can also participate in the telephone survey through interpretors. Only one adult in each household that is contacted can complete the survey. Of all potential survey respondents, about one-half will provide complete data for the telephone survey.
Sampling Method: Non-Probability Sample
Enrollment: 40690 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of persons with or at high-risk of COPD | 1 year
  COPD defined by respondent self-report; high-risk for COPD defined by frequency of respiratory symptoms and tobacco exposure history

SECONDARY OUTCOMES:
Prevalence of respiratory symptoms in general adult population | 1 year
  Telephone health survey using the Behavioral Risk factor Surveillance System to define the frequency of dyspnea
Relationship between racial and socioeconomic disparities with respiratory symptoms | 1 year
  Telephone health survey using the Behavioral Risk Factor Surveillance System to define the frequency of respiratory symptoms (%) based upon respondent's race, ethnicity (Hispanic, non-Hispanic), annual income ($), educational status (< high school, HS, some college, college graduate) with frequency (%) and severity of respiratory symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Njira Lugogo, MD, Study Director — Duke University

IPD SHARING:
Plan to Share IPD: Yes
Through respective state's BRFSS